CLINICAL TRIAL: NCT00883428
Title: Prevalence of Low Back and Pelvic Pain in Pregnant Women and Factors Associated With a Greater Risk of Having it
Brief Title: Prevalence of Low Back and Pelvic Pain in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK 28
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Low Back Pain; Pelvic Pain
Keywords: low back pain; pelvic pain; pregnancy
MeSH Terms: conditions — Low Back Pain; Pelvic Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pergnant women: Pregnant women, of 28 weeks or more of gestation, who are seen in the Health Centers participating in the study.
  Interventions: Other: Set of questionnaires

INTERVENTIONS:
Other: Set of questionnaires — A set of questionnaires to determine the existence of low back and pelvic pain during the pregnancy, and to identify possible risk factors.

SUMMARY:
The purpose of this study is to determine the prevalence of low back and pelvic pain in Spanish pregnant women. The results should allow for the identification of factors associated with a greater risk of having it during pregnancy. Once risk factors are identified, other studies can assess the effectiveness of measures to reduce this pain.

DETAILED DESCRIPTION:
Validated methods were used to gather data on the prevalence of LBP, LP and PGP, anthropometric and socio-demographic characteristics, history of LBP, obstetrical history, physical activity before and during pregnancy, mattress and sleep characteristics, disability, anxiety, and depression. Separate multiple logistic regression models were developed to identify the variables associated with LBP, LP and PGP.

ELIGIBILITY:
Inclusion Criteria:

* A pregnancy of 28 weeks or more
* Able to understand, read and write Spanish
* Seen at participating health centers or hospitals in the study
* Signs informed consent form

Exclusion Criteria:

* Refusal to participate in the study
* Being under 18 years of age or legally mentally incapacitated
* Having a diagnosis of illnesses that can cause back pain

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who are 28 weeks pregnant or more (in the third trimester of the pregnancy).
Sampling Method: Non-Probability Sample
Enrollment: 1158 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The prevalence of low back and pelvic pain in pregnant women, measured in the third trimester of pregnancy. | 24 months

SECONDARY OUTCOMES:
The influence of risk factors, such as anxiety or depression, on low back and pelvic pain in pregnant women. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Betina Nishishinya, MD, Principal Investigator — Kovacs Foundation, Palma de Mallorca, 07012, Spain
Locations (20):
- Spain (20):
  - Centro de Salud de Ciudad Jardín, Málaga, Andalusia
  - Centro de Salud El Limonar, Málaga, Andalusia
  - Centro de Salud de Andratx, Andraxt, Balearic Islands
  - Centro de Salud de Campos, Campos, Balearic Islands
  - Centro de Salud Lluchmajor - Mitjorn, Lluchmajor, Balearic Islands
  - Centro de Salud de La Vileta, Palma de Mallorca, Balearic Islands
  - Centro de Salud del Col dén Rabassa, Palma de Mallorca, Balearic Islands
  - Centro de Salud del Rafal Nou, Palma de Mallorca, Balearic Islands
  - Centro de Salud Son Rullán, Palma de Mallorca, Balearic Islands
  - Centro de Salud del Campo Redó, Palma de Mallorca, Balearic Islands
  - Centro de Salud de Son Pisá, Palma de Mallorca, Balearic Islands
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Kovacs Foundation, Palma de Mallorca, Balearic Islands
  - Centro de Salud de Santa Catalina, Palma de Mallorca, Balearic Islands
  - Centro de Salud de Valldargent, Palma de Mallorca, Balearic Islands
  - Centro de Salud de Santa Ponsa, Santa Ponsa, Balearic Islands
  - Centro de Salud de Bembibre, Bembibre, León
  - Depto. de Enfermería y Fisioterapia, Universidad de León, Ponferrada, León
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Centro de Salud Benita de Avila, Madrid, Madrid

REFERENCES:
- [Background] Fast A, Shapiro D, Ducommun EJ, Friedmann LW, Bouklas T, Floman Y. Low-back pain in pregnancy. Spine (Phila Pa 1976). 1987 May;12(4):368-71. doi: 10.1097/00007632-198705000-00011. PMID 2956698
- [Background] Mens JM, Vleeming A, Stoeckart R, Stam HJ, Snijders CJ. Understanding peripartum pelvic pain. Implications of a patient survey. Spine (Phila Pa 1976). 1996 Jun 1;21(11):1363-9; discussion 1369-70. doi: 10.1097/00007632-199606010-00017. PMID 8725930
- [Background] Orvieto R, Achiron A, Ben-Rafael Z, Gelernter I, Achiron R. Low-back pain of pregnancy. Acta Obstet Gynecol Scand. 1994 Mar;73(3):209-14. doi: 10.3109/00016349409023441. PMID 8122500